CLINICAL TRIAL: NCT06753084
Title: Keratinized Tissue Augmentation Using Porcine Collagen Matrix (Mucoderm®) Around Dental Implant: A Randomized Clinical Study
Brief Title: Keratinized Tissue Augmentation Using Porcine Collagen Matrix (Mucoderm®) Around Dental Implant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ahmed amer (Other)
Collaborators: Misr University for Science and Technology (Other)
Responsible Party: Sponsor-Investigator, ahmed amer, teaching assistant periodontics department faculty of dentistry, Misr University for Science and Technology
Organization: Misr University for Science and Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KTW Managment
Record Dates: First submitted 2024-12-16; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Keratinized Mucosa
Keywords: keratinized tissue width , porcine collagen matrix
MeSH Terms: interventions — Alloderm

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- KTW augmentation using FGG (Active Comparator): KTW augmentation using apically positioned flap combined with FGG from palatal mucosa
  Interventions: Procedure: Alloderm
- KTW augmentation using porcine collagen matrix (Experimental): KTW augmentation using apically positioned flap combined with porcine collagen matrix
  Interventions: Procedure: Alloderm

INTERVENTIONS:
Procedure: Alloderm — the study is done to patient who lacks of keratinized mucosa width by apically positioned flap and using of FGG as gold standard and Mucoderm as compartive group

SUMMARY:
Aim of the Study To evaluate the using of porcine collagen matrix for keratinized tissue augmentation around delayed dental implant.

Primary Outcome:

Peri-implant keratinized mucosal width and thickness following the use of porcine collagen matrix using (Mucoderm®-Botiss gmbh) compared to the gold standard FGG augmentation.

Secondary Outcome:

1. Crestal bone change (CBC)
2. Pocket depth (PD)
3. Bleeding on probing (BOP)
4. Plaque index (PI) PICOT

P: Population:

Patient with suitable ridge dimension for delayed implant placement.

I: Intervention:

Implant insertion followed by porcine collagen matrix soft tissue augmentation

C: Control:

Autogenous FGG

O: Outcomes

* Enhancing keratinized mucosal width and thickness
* Evaluating :

  1. Crestal bone change (CBC)
  2. perimplant Pocket depth (PD)
  3. Bleeding on probing (BOP)
  4. Plaque index (PI)
  5. Modified PES. T: Time A 6 months follow up .

DETAILED DESCRIPTION:
this study aiming to augment KMW with FGG and MUCODERM following apically positioned flap the primary outcomes to measure is KMW and MT

ELIGIBILITY:
Inclusion Criteria:

* 1- Partially or fully edentulous sites with previous implant placed in posterior maxillary or mandibular areas.

  2- Inadequate keratinized tissue ≤2 3- Patient age ranged from 20 to 45 years old for both genders. 4- Submerged Osteointegrated implants with no sings of inflammation before implant insertion.

  5- Optimal compliance as evidenced by no missed treatment appointments and positive attitude toward oral hygiene.

Exclusion Criteria:

* 1- Smokers 2- Pregnant or lactating female 3- Treatment with any systemic drug that could affect wound healing (ex- corticosteroids ) 4- History of systemic disease affect wound healing ex diabetes 5- Patient with bruxism and parafunctional habits. 6- Limited inter arch restoration space.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Keratinized mucosa width | 1 month , 3 month , 6 months follow up
  before the operation reading , immediately after operation , 1 month follow up , 3 months follow up and 6 months follow up
  the reading will done using periodontal probe
keratinized tissue thickness | 1 month , 3 month , 6 months follow up
  measures the Keratinized tissue thickness using periodontal probe

SECONDARY OUTCOMES:
probing depth for adjacent teeth | 6 months
  probing depth for adjacent teeth
bleeding on probingn | 1 month , 3 month , 6 months follow up
  bleeding on probing for this patient is mesure using papillary bleeding index.
crestal bone loss around dental implant | 1 month , 3 month , 6 months follow up
  measuring crestal bone loss around implant using CBCT and periapical xray

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Misr university for science and technology, Giza, NJ
  - Misr university for science and technology, Giza

IPD SHARING:
Plan to Share IPD: Undecided
after thesis discussion we will decide